CLINICAL TRIAL: NCT03779542
Title: Assessment Of Anterior Chamber Configuration Changes After Phacoemulsification With Swept-Source Optical Coherence Tomography
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Yune Zhao (Other)
Responsible Party: Sponsor-Investigator, Yune Zhao, Director, Wenzhou Medical University
Organization: Wenzhou Medical University (Other)
Other Study IDs: HM-AOD-HZ
Record Dates: First submitted 2018-12-17; First posted 2018-12-19 (Actual); Last update posted 2018-12-19 (Actual); Status verified 2018-12

CONDITIONS: Anterior Chamber Parameters; Phacoemulsification; Anterior Segment Swept-source Optical Coherence Tomography
Keywords: anterior chamber parameters; phacoemulsification; anterior segment swept-source optical coherence tomography
MeSH Terms: interventions — Cataract Extraction

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- open-angle group: ACD > 2.68 measured by the swept source AS-OCT and angle > Shaffer 2 in four quadrants under gonioscope
  Interventions: Procedure: cataract surgery
- narrow-angle group: ACD≤2.68 measured by the swept source AS-OCT and angle≤Shaffer 2 in four quadrants under gonioscope
  Interventions: Procedure: cataract surgery

INTERVENTIONS:
Procedure: cataract surgery — phacoemulsification and intraocular lens implantation

SUMMARY:
To assess the changes of anterior chamber angle in patients with shallow anterior chamber and normal anterior chamber after phacoemulsification and intraocular lens implantation (IOL) using anterior segment swept-source optical coherence tomography (AS-SS-OCT).To observe the 60 eyes of 60 patients in our study.

DETAILED DESCRIPTION:
This is a prospective case-control study; 60 eyes of 60 patients who underwent cataract surgery. Based on anterior chamber depth (ACD) and gonioscopy findings, the eyes are classified into two groups, shallow anterior chamber group (30 eyes) and narrow anterior chamber group (30 eyes). AS-SS-OCT was used to measure ACD and angle parameters (angle opening distance(AOD), angle recess area(ARA), trabecular iris space area（TISA）, and trabecular iris angle (TIA). Serial changes in each group were measured before and 3 months after phacoemulsification and IOL, and the differences between the two groups were compared.

ELIGIBILITY:
Inclusion Criteria: patients who underwent cataract surgery -

Exclusion Criteria:patients with mild cataracts do not require surgery

-

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients who underwent cataract surgery
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2018-01-01 (Actual); Primary Completion 2018-06-30 (Actual); Study Completion 2019-06 (Estimated)

PRIMARY OUTCOMES:
anterior chamber depth | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Eye Hospital of Wenzhou Medical College, Wenzhou, Zhejiang, China